CLINICAL TRIAL: NCT01376700
Title: A Phase 3b Clinical Study to Assess Whether Regular Administration of ADVATE in the Absence of Immunological Danger Signals Reduces the Incidence Rate of Inhibitors in Previously Untreated Patients With Hemophilia A
Brief Title: Early Prophylaxis Immunologic Challenge (EPIC) Study
Acronym: EPIC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: It became unlikely to achieve the study objective of 50% reduction over published inhibitor rates. The Data Monitoring Committee supported this decision.
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Baxter Innovations GmbH (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 061002; 2011-000410-18 (EudraCT Number)
Record Dates: First submitted 2011-06-17; First posted 2011-06-20 (Estimated); Results first posted 2014-10-09 (Estimated); Last update posted 2021-05-24 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ADVATE - Prophylactic Regimen (Experimental): Weekly infusions of ADVATE. Study visits (physical examination, lab tests including FVIII inhibitor tests) every week during the first 10 exposure days (EDs), every 5 weeks during the next 10 EDs and every 10 weeks thereafter.
  Interventions: Biological: Recombinant antihemophilic factor, plasma/albumin-free method (rAHF-PFM)

INTERVENTIONS:
Biological: Recombinant antihemophilic factor, plasma/albumin-free method (rAHF-PFM) — Intravenous infusion at a dose of 25 ± 5 IU/kg once per week. After 20 exposure days, the weekly infusions should be continued for as long as possible following the early prophylaxis period. If required by the clinical situation, dosing may be increased to twice weekly or even three times weekly after 20 exposure days, while keeping the low dose.
  Other Names: ADVATE

SUMMARY:
The purpose of the study was to assess if a once-weekly prophylactic regimen of 25 IU/kg ADVATE started at or before 1 year of age and before the onset of a severe bleeding phenotype (ie, joint bleeding), together with the minimization of immunological danger signals, can reduce the incidence rate of inhibitor formation in PUPs with severe and moderately severe hemophilia A.

ELIGIBILITY:
Inclusion Criteria:

* Participants with severe and moderately severe hemophilia A (FVIII ≤ 2%)
* Participants < 1 year of age
* Participants must have ≤ 3 exposure days (EDs) to any FVIII concentrate or FVIII-containing product used for treatment of minor bleeds (bleeds requiring no more than 2 infusions per event), or for preventative or precautionary infusions following possible injury
* Participants with prior circumcision are allowed to enroll only if bleeding issues related to circumcision were the cause for the original diagnosis of hemophilia A and no more than 2 EDs of FVIII treatment were required
* Adequate venous access (without need for central venous access device (CVAD)-placement) as determined by the physician
* Written informed consent from legally authorized representative(s)

Exclusion Criteria:

* Life-threatening conditions (intracranial hemorrhage, severe trauma) or requirement for surgery at the time of enrollment
* Evidence of inhibitor ≥ 0.6 Bethesda Unit (BU) in Nijmegen-modified Bethesda Assay at study start (samples may be retested using lupus-insensitive inhibitor tests to reduce the number of false positive inhibitor test results)
* Inherited or acquired hemostatic defect other than hemophilia A
* Any clinically significant, chronic disease other than hemophilia A
* Known hypersensitivity to ADVATE or any of its constituents
* Any planned elective surgery that cannot be postponed until after the first 20 EDs
* Participation in the Hemophilia Inhibitor Previously Untreated Patient Study
* Application of red blood cell, platelet, or leukocyte concentrates, or plasma
* Administration of any medication affecting coagulation or platelet function
* Systemic administration of any immunomodulatory drug (eg, chemotherapy, intravenous glucocorticoids)
* Participation in another clinical study involving an investigational product (IP) or device within 30 days prior to study enrollment or during the course of this study

Max Age: 1 Year | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2011-08-26 (Actual); Primary Completion 2012-11-16 (Actual); Study Completion 2012-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (19):
- United States (2):
  - Indianapolis, Indiana
  - New Brunswick, New Jersey
- Vienna, Austria
- Sofia, Bulgaria
- Kingston, Ontario, Canada
- Brno, Czechia
- Germany (4):
  - Bonn
  - Bremen
  - Giessen
  - Munich
- Vilnius, Lithuania
- Nijmegen, Netherlands
- Poland (2):
  - Lublin
  - Olsztyn
- Russia (3):
  - Chelyabinsk
  - Krasnodar
  - Saint Petersburg
- Belgrade, Serbia
- A Coruña, Spain

REFERENCES:
- [Result] Auerswald G, Kurnik K, Aledort LM, Chehadeh H, Loew-Baselli A, Steinitz K, Reininger AJ; EPIC clinical study group. The EPIC study: a lesson to learn. Haemophilia. 2015 Sep;21(5):622-8. doi: 10.1111/hae.12666. Epub 2015 Apr 23. PMID 25912619

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was conducted in Europe and North America at 19 clinical sites.
Pre-assignment Details: 22 participants were enrolled. One was a screen failure; one did not have screening laboratory assessments performed prior to study termination; and one met screening criteria, but was not exposed to investigational product prior to study termination. Therefore 19 participants were treated
Period: Overall Study
Arm/Group | ADVATE - Prophylactic Regimen
Started | 19
Completed | 3
Not Completed | 16
Not completed — Sponsor terminated study early | 8
Not completed — Low or high titer inhibitor | 8

BASELINE CHARACTERISTICS:
Arm/Group | ADVATE - Prophylactic Regimen
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 43.3 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 19
Region of Enrollment [Count of Participants; unit: Participants]
  Serbia | 1
  United States | 2
  Czech Republic | 2
  Canada | 1
  Spain | 1
  Poland | 4
  Austria | 1
  Russian Federation | 3
  Bulgaria | 1
  Netherlands | 1
  Germany | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Severe and Moderately Severe Hemophilia A (FVIII ≤ 2%) With Factor VIII (FVIII) Inhibitor Formation Within the First 50 Exposure Days to ADVATE
Description: Inhibitor testing will be performed in the central laboratory and a non-zero result must be confirmed in the central laboratory as soon as possible, preferably 1 week after inhibitor testing. Confirmed FVIII inhibitor is defined as any FVIII inhibitor assay result equal or greater than 0.6 Bethesda Units (BU)/mL confirmed by the central laboratory on 2 consecutive samples, i.e. at least 2 positive inhibitor results (including the first positive inhibitor test, in accordance with the study protocol) assessed as either: - i. High FVIII inhibitor titer (> 5 BU/mL) or - ii. Low FVIII inhibitor titer (≥0.6 - ≤5.0 BU/mL).
Time Frame: 50 exposure days to ADVATE
Population: Safety Analysis Set All study participants had severe Hemophilia A, less than 1% Factor VIII levels. (ie there were no moderately severe hemophilia A participants (FVIII levels >1% to ≤ 2%) in this study.
Measure: Number; unit: participants
Groups:
- ADVATE - Prophylactic Regimen: Weekly infusions of ADVATE. Study visits (physical examination, lab tests including FVIII inhibitor tests) every week during the first 10 exposure days (EDs), every 5 weeks during the next 10 EDs and every 10 weeks thereafter. Recombinant antihemophilic factor, plasma/albumin-free method (rAHF-PFM): Intravenous infusion at a dose of 25 ± 5 IU/kg once per week. After 20 exposure days, the weekly infusions should be continued for as long as possible following the early prophylaxis period. If required by the clinical situation, dosing may be increased to twice weekly or even three times weekly after 20 exposure days, while keeping the low dose.
Arm/Group | ADVATE - Prophylactic Regimen
Number analyzed (Participants) | 19
participants | 8

2. Secondary Outcome: Number of Participants With Severe Hemophilia A (FVIII ≤ 1%) With Factor VIII (FVIII) Inhibitor Formation Within the First 50 Exposure Days to ADVATE
Description: as for outcome 1
Time Frame: 50 exposure days to ADVATE
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | ADVATE - Prophylactic Regimen
Number analyzed (Participants) | 19
participants | 8

3. Secondary Outcome: Number of Exposure Days of Treatment With Advate Prior to First Positive Factor VIII (FVIII) Confirmed Inhibitor Assessment
Description: Confirmed inhibitor is defined as any FVIII inhibitor assay result equal or greater than 0.6 BU/mL confirmed by the central laboratory on 2 consecutive samples, i.e. at least 2 positive inhibitor results (including the first positive inhibitor test, in accordance with the study protocol) assessed as either: - i. High FVIII inhibitor titer (> 5 BU/mL) or - ii. Low FVIII inhibitor titer (≥0.6 - ≤5.0 BU/mL).
Time Frame: 50 exposure days to ADVATE
Population: Safety Analysis Set
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | ADVATE - Prophylactic Regimen
Number analyzed (Participants) | 19
days | 14.5 [7.0 to 21.0]

4. Secondary Outcome: Number of Participants With Low-titer, High-titer, Transient, and All Factor VIII (FVIII) Inhibitors
Description: - High FVIII inhibitor titer (> 5 Bethesda Unit (BU)/mL) - Low FVIII inhibitor titer (≥0.6 - ≤5.0 BU/mL)
Time Frame: 50 exposure days to ADVATE
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | ADVATE - Prophylactic Regimen
Number analyzed (Participants) | 19
participants
  Low FVIII inhibitor titer | 5
  High FVIII inhibitor titer | 3
  All FVIII inhibitors | 8

5. Secondary Outcome: Number, Type, and Severity of All Bleeds Experienced When Different Prophylactic Dosing Frequencies Are Used (Once or Twice Per Week and Unknown Frequency)
Description: Nominal Dosing Frequency: - 1 time per week - 2 times per week - Unknown dosing frequency (UK) Bleeding Type (BT): - Skin - Muscle and Soft Tissue - Mucosal - Joint - Other - Multiple - Total Bleeding severity: - Minor - Moderate - Severe - Total
Time Frame: 50 exposure days to ADVATE
Population: Safety Analysis Set
Measure: Number; unit: Bleeds
Units Other Than Participants: Bleeds
Arm/Group | ADVATE - Prophylactic Regimen
Number analyzed (Participants) | 19
Number analyzed (Bleeds) | 193
Bleeds
  Dose: 1/week; Skin; Minor Bleed | 130
  Dose: 1/week; Skin; Moderate Bleed | 2
  Dose: 1/week; Skin; Severe Bleed | 0
  Dose: 1/week; Skin; Total Bleeds | 132
  Dose: 1/week; Muscle & Soft Tissue; Minor Bleed | 8
  Dose: 1/week; Muscle & Soft Tissue; Moderate Bleed | 10
  Dose: 1/week; Muscle & Soft Tissue; Severe Bleed | 0
  Dose: 1/week; Muscle & Soft Tissue; Total Bleeds | 18
  Dose: 1/week; Mucosal; Minor Bleed | 9
  Dose: 1/week; Mucosal; Moderate Bleed | 3
  Dose: 1/week; Mucosal; Severe Bleed | 0
  Dose: 1/week; Mucosal; Total Bleeds | 12
  Dose: 1/week; Joint; Minor Bleed | 0
  Dose: 1/week; Joint; Moderate Bleed | 0
  Dose: 1/week; Joint; Severe Bleed | 0
  Dose: 1/week; Joint; Total Bleeds | 0
  Dose: 1/week; Other BT; Minor Bleed | 3
  Dose: 1/week; Other BT; Moderate Bleed | 3
  Dose: 1/week; Other BT; Severe Bleed | 1
  Dose: 1/week; Other BT; Total Bleeds | 7
  Dose: 1/week; Multiple BT; Minor Bleed | 2
  Dose: 1/week; Multiple BT; Moderate Bleed | 1
  Dose: 1/week; Multiple BT; Severe Bleed | 0
  Dose: 1/week; Multiple BT; Total Bleeds | 3
  Dose: 1/week; Total BT; Minor Bleed | 152
  Dose: 1/week; Total BT; Moderate Bleed | 19
  Dose: 1/week; Total BT; Severe Bleed | 1
  Dose: 1/week; Total BT; Total Bleeds | 172
  Dose: 2/week; Skin; Minor Bleed | 9
  Dose: 2/week; Skin; Moderate Bleed | 0
  Dose: 2/week; Skin; Severe Bleed | 0
  Dose: 2/week; Skin; Total Bleeds | 9
  Dose: 2/week; Muscle & Soft Tissue; Minor Bleed | 0
  Dose: 2/week; Muscle & Soft Tissue; Moderate Bleed | 1
  Dose: 2/week; Muscle & Soft Tissue; Severe Bleed | 0
  Dose: 2/week; Muscle & Soft Tissue; Total Bleeds | 1
  Dose: 2/week; Mucosal; Minor Bleed | 3
  Dose: 2/week; Mucosal; Moderate Bleed | 1
  Dose: 2/week; Mucosal; Severe Bleed | 0
  Dose: 2/week; Mucosal; Total Bleeds | 4
  Dose: 2/week; Joint; Minor Bleed | 0
  Dose: 2/week; Joint; Moderate Bleed | 0
  Dose: 2/week; Joint; Severe Bleed | 0
  Dose: 2/week; Joint; Total Bleeds | 0
  Dose: 2/week; Other BT; Minor Bleed | 0
  Dose: 2/week; Other BT; Moderate Bleed | 0
  Dose: 2/week; Other BT; Severe Bleed | 0
  Dose: 2/week; Other BT; Total Bleeds | 0
  Dose: 2/week; Multiple BT; Minor Bleed | 0
  Dose: 2/week; Multiple BT; Moderate Bleed | 0
  Dose: 2/week; Multiple BT; Severe Bleed | 0
  Dose: 2/week; Multiple BT; Total Bleeds | 0
  Dose: 2/week; Total BT; Minor Bleed | 12
  Dose: 2/week; Total BT; Moderate Bleed | 2
  Dose: 2/week; Total BT; Severe Bleed | 0
  Dose: 2/week; Total BT; Total Bleeds | 14
  Dose: UK/week; Skin; Minor Bleed | 4
  Dose: UK/week; Skin; Moderate Bleed | 1
  Dose: UK/week; Skin; Severe Bleed | 0
  Dose: UK/week; Skin; Total Bleeds | 5
  Dose: UK/week; Muscle & Soft Tissue; Minor Bleed | 0
  Dose: UK/week; Muscle & Soft Tissue;Moderate Bleed | 1
  Dose: UK/week; Muscle & Soft Tissue; Severe Bleed | 0
  Dose: UK/week; Muscle & Soft Tissue; Total Bleeds | 1
  Dose: UK/week; Mucosal; Minor Bleed | 0
  Dose: UK/week; Mucosal; Moderate Bleed | 0
  Dose: UK/week; Mucosal; Severe Bleed | 0
  Dose: UK/week; Mucosal; Total Bleeds | 0
  Dose: UK/week; Joint; Minor Bleed | 0
  Dose: UK/week; Joint; Moderate Bleed | 1
  Dose: UK/week; Joint; Severe Bleed | 0
  Dose: UK/week; Joint; Total Bleeds | 1
  Dose: UK/week; Other BT; Minor Bleed | 0
  Dose: UK/week; Other BT; Moderate Bleed | 0
  Dose: UK/week; Other BT; Severe Bleed | 0
  Dose: UK/week; Other BT; Total Bleeds | 0
  Dose: UK/week; Multiple BT; Minor Bleed | 0
  Dose: UK/week; Multiple BT; Moderate Bleed | 0
  Dose: UK /week; Multiple BT; Severe Bleed | 0
  Dose: UK /week; Multiple BT; Total Bleeds | 0
  Dose: UK /week; Total BT; Minor Bleed | 4
  Dose: UK /week; Total BT; Moderate Bleed | 3
  Dose: UK /week; Total BT; Severe Bleed | 0
  Dose: UK /week; Total BT; Total Bleeds | 7

6. Secondary Outcome: Number and Type of Surgeries
Description: - Elective surgery is not allowed during period of first 20 exposure days (EDs) - Peripherally inserted central catheter (PICC)
Time Frame: 50 exposure days to ADVATE
Population: Safety Analysis Set
Measure: Number; unit: surgeries
Arm/Group | ADVATE - Prophylactic Regimen
Number analyzed (Participants) | 19
surgeries
  Surgery: Cimino Shunt | 1
  Surgery: PICC Line Insertion in right arm | 1

7. Secondary Outcome: Correlation of Known Risk Factors to Factor VIII (FVIII) Inhibitor Formation
Time Frame: 50 exposure days to ADVATE
Population: Due to the low number of subjects available for evaluation, no statistical tests were performed to assess associations between known risk factors to inhibitor formation.
Arm/Group | ADVATE - Prophylactic Regimen
Number analyzed (Participants) | 0

8. Secondary Outcome: Total Factor VIII (FVIII) Consumption by Participant
Time Frame: 50 exposure days to ADVATE
Population: Due to the low number of subjects available for evaluation, no statistical tests were performed to assess the total FVIII consumption by participant
Arm/Group | ADVATE - Prophylactic Regimen
Number analyzed (Participants) | 0

9. Secondary Outcome: FVIII-Specific Antibody Isotype for All Participants at Study Entry and Every 10 Exposure Days (EDs)
Time Frame: 50 exposure days to ADVATE
Population: Summary statistics of FVIII-Specific Antibody Isotypes were not performed due to the early termination of the study
Arm/Group | ADVATE - Prophylactic Regimen
Number analyzed (Participants) | 0

10. Secondary Outcome: Number of Serious Adverse Events (SAEs) and Non-serious Adverse Events (Non-SAEs) at Least Possibly Related to ADVATE
Description: Possibly or probably related adverse events
Time Frame: 50 exposure days to ADVATE
Population: Safety Analysis Set
Measure: Number; unit: adverse events
Arm/Group | ADVATE - Prophylactic Regimen
Number analyzed (Participants) | 19
adverse events
  SAEs | 9
  non-SAEs | 1

11. Post Hoc Outcome: Number of Participants With Factor VIII (FVIII) Inhibitors by Inhibitor Type (Only 'True' Inhibitors)
Description: 'True' positive inhibitor (PI) defined as any FVIII inhibitor assay result ≥0.6 Bethesda Units (BU)/mL confirmed by central lab on 2 consecutive samples, ie ≥2 PI results (including first PI test, in accordance with study protocol) assessed as either: i. High FVIII inhibitor titer (> 5 BU/mL) ii. Low FVIII inhibitor titer (≥0.6 - ≤5.0 BU/mL). In addition, to be classified as 'true' positive low FVIII inhibitors titer (≥0.6 - ≤5.0 BU/mL), one of following criteria must be met: - a) Lower or absent therapeutic response at infusion of standard replacement doses ("clinically relevant") as deemed by the clinician in charge. - b) Any lab result of binding FVIII antibodies (IgM, IgA, IgG, IgG1, IgG2, IgG3, or IgG4) must be positive. Classification based on first positive FVIII inhibitor assessment. Inhibitor test result is: - > 5 BU/mL, then categorized as a high-titer inhibitor - ≥0.6 BU/mL but ≤5 BU/mL, then categorized as a low-titer.
Time Frame: 50 exposure days to ADVATE
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | ADVATE - Prophylactic Regimen
Number analyzed (Participants) | 19
participants
  Inhibitor Type: Low-Titer | 3 [3.4 to 39.6]
  Inhibitor Type: High-Titer | 3 [3.4 to 39.6]
  Inhibitor Type: All Inhibitors | 6 [12.6 to 56.6]

12. Post Hoc Outcome: Number of Inhibitors in Previously Untreated Patients (PUPs) and Minimally Treated Patients (MTPs) - (Only 'True' Inhibitors)
Description: PUPs = no previous FVIII exposure; MTPs ≤4 previous FVIII exposures 'True' positive inhibitor (PI) = any FVIII inhibitor assay result ≥0.6 Bethesda Units (BU)/mL confirmed by central lab on 2 consecutive samples, ie ≥2 PI results (including first PI test, per study protocol) assessed as either: i. High FVIII inhibitor titer (>5 BU/mL) ii. Low FVIII inhibitor titer (≥0.6 - ≤5.0 BU/mL). In addition, to be classified as 'true' positive low FVIII inhibitors titer (≥0.6 - ≤5.0 BU/mL), one of following criteria must be met: - a) Lower or absent therapeutic response at infusion of standard replacement doses ("clinically relevant") as deemed by clinician in charge. - b) Any lab result of binding FVIII antibodies (IgM, IgA, IgG, IgG1, IgG2, IgG3, or IgG4) must be positive. Classification based on first positive FVIII inhibitor assessment. Inhibitor test result is: - > 5 BU/mL, categorized as high-titer inhibitor - ≥0.6 BU/mL but ≤5 BU/mL, categorized as low-titer
Time Frame: 50 exposure days to ADVATE
Population: Safety Analysis Set
Measure: Number; unit: inhibitors
Groups:
- PUPs: No previous FVIII exposure
- MTPs: ≤4 previous FVIII exposures
Arm/Group | PUPs | MTPs
Number analyzed (Participants) | 11 | 8
inhibitors | 3 | 3

ADVERSE EVENTS:
Time Frame: 1 year and 3 months
Arm/Group | ADVATE - Prophylactic Regimen
Serious Adverse Events (participants affected / at risk) | 11/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADVATE - Prophylactic Regimen (N=19)
FACTOR VIII INHIBITION (Blood and lymphatic system disorders) | 8 (8)
HEAD INJURY (Injury, poisoning and procedural complications) | 1 (1)
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 1 (2)
SOFT TISSUE HAEMORRHAGE (Musculoskeletal and connective tissue disorders) | 1 (1)
ARTERIOVENOUS FISTULA OPERATION (Surgical and medical procedures) | 1 (1)
HAEMORRHAGE (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADVATE - Prophylactic Regimen (N=19)
FACTOR VIII INHIBITION (UNCONFIRMED) (Blood and lymphatic system disorders) | 1 (1)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 (1)
MIDDLE EAR EFFUSION (Ear and labyrinth disorders) | 1 (1)
EYE DISCHARGE (Eye disorders) | 1 (1)
LACRIMATION INCREASED (Eye disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 3 (3)
TEETHING (Gastrointestinal disorders) | 4 (10)
VOMITING (Gastrointestinal disorders) | 5 (6)
PYREXIA (General disorders) | 10 (13)
FOOD ALLERGY (Immune system disorders) | 1 (1)
ACUTE TONSILLITIS (Infections and infestations) | 1 (2)
BRONCHITIS (Infections and infestations) | 1 (2)
CANDIDIASIS (Infections and infestations) | 1 (1)
COXSACKIE VIRAL INFECTION (Infections and infestations) | 1 (1)
EAR INFECTION (Infections and infestations) | 2 (2)
GASTROENTERITIS (Infections and infestations) | 1 (2)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1)
HORDEOLUM (Infections and infestations) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 6 (7)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1)
RHINITIS (Infections and infestations) | 8 (13)
TONSILLITIS (Infections and infestations) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (7)
VIRAL INFECTION (Infections and infestations) | 1 (1)
FACE INJURY (Injury, poisoning and procedural complications) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1)
LIP INJURY (Injury, poisoning and procedural complications) | 1 (2)
TONGUE INJURY (Injury, poisoning and procedural complications) | 1 (1)
VACCINATION COMPLICATION (Injury, poisoning and procedural complications) | 1 (1)
WRONG DRUG ADMINISTERED (Injury, poisoning and procedural complications) | 1 (3)
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 1 (1)
JOINT RANGE OF MOTION DECREASED (Musculoskeletal and connective tissue disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 (6)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 1 (2)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 2 (3)
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 (1)
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 1 (1)
DERMATITIS DIAPER (Skin and subcutaneous tissue disorders) | 1 (5)
ECZEMA (Skin and subcutaneous tissue disorders) | 1 (1)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 3 (3)
HAEMATOMA (Vascular disorders) | 1 (1)
VASCULAR RUPTURE (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination lead to: -No statistical tests done on risk factors & inhibitor formation. -FVIII consumption by participant not calculated due to large variation in # of EDs. -FVIII-Specific Antibody Isotypes summary statistics not done.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreements may vary with individual PIs, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication or up to 2 years after study completion. Baxter requires a review of results communications (eg for confidential information) ≥30 days prior to submission/communication. Baxter may request additional delay of ≤6 months (e.g., for intellectual property protection). Prior authorization may be required